CLINICAL TRIAL: NCT06852833
Title: One-day Mind Programme for Women With Breast Cancer: A Pilot Study on the Acceptability and Effectiveness of a Brief ACT and Compassion-based Intervention on Breast Cancer-specific Outcomes
Brief Title: One-day Mind Programme for Women With Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Portuguese National Funding Agency for Science, Research and Technology (FCT) (Unknown)
Responsible Party: Principal Investigator, Inês A Trindade, CINEICC Collaborative member, University of Coimbra
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINEICC-3-IAT(brief); PTDC/PSI-GER/7847/2020 (Other Grant/Funding Number: Fundação para a Ciência e a Tecnologia, I.P./MCTES)
Record Dates: First submitted 2025-02-10; First posted 2025-02-28 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Females
Keywords: Breast Cancer; Contextual Behavioural Therapies; Psychological Flexibility; Self-compassion; Cancer-related Quality of Life; Mental Health; ACT; Psycho-oncology; Oncology; Women; Brief Psychological Intervention
MeSH Terms: conditions — Breast Neoplasms; Psychological Well-Being; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mind (brief) (Experimental): This group will receive the "One-day Mind Programme for women with breast cancer" (see description in the next box) in two different days. All participants will continue on receiving the recommended medical treatment for their clinical diagnosis.
  Interventions: Behavioral: One-day Mind Programme for women with breast cancer

INTERVENTIONS:
Behavioral: One-day Mind Programme for women with breast cancer — This programme is theoretically founded on contextual behavioural therapies ( ACT and compassion-based interventions) and tailored for women with breast cancer. Its format comprises 1 session with the duration of 7 hours, that will be delivered by 2 psychologists through a secure video calling platform, in two subsequent days.

SUMMARY:
Breast cancer (BC) remains the second most common type of cancer worldwide and the leading cancer affecting women. In Portugal there are approximately 7000 new diagnoses of BC each year. The diagnosis and treatment of BC can profoundly impact patients' physical (e.g., fatigue, pain) and psychological (e.g. distress, depressive symptoms) well-being. Psychological interventions that foster adjustment to cancer (and to its treatment), mental health and quality of life are therefore essential.

The use of contextual behavioural therapies in samples of people with chronic diseases has shown evidence of efficacy in improving psychopathological symptoms. Additionally, a recent meta-analysis concluded that the use of single-session ACT interventions in samples with chronically ill patients may be more viable, acceptable, and beneficial compared to multiple-session ACT interventions.

This interventional study aims to test the acceptability (aim 1) and effectiveness (aim 2) of a brief (7-hour) version of the "Mind Programme for Women with Breast Cancer", which is providing promising efficacy results. Similarly to the original programme, this brief version integrates contextual behavioural therapies (Acceptance and Commitment Therapy - ACT, and Compassion-Focused Therapy - CFT), is tailored to BC women and presents a group and online format, delivered by two psychologists. This trial also aims to determine the contribution of mediating (psychological flexibility, self-compassion) and moderating (e.g. age) factors in treatment effectiveness (aim 3).

Women with BC who had previously shown interest in participating in the RCT of the (original) multiple-session Mind Programme, but that were either not eligible or were allocated to the waiting list, will be invited to join this trial. Participants will complete the 7-h intervention "One-day Mind Programme for women with breast cancer" and complete self-reported outcome measures (e.g. EORTC QLQ-C30, HADS, CompACT, SCS, resource use questionnaire) in three different timepoints (pre, post, and 3-month follow-up). The G*Power 3.1.9.7 software was used to calculate the sample size (N=36) required for a single-armed linear repeated-measures model with three measurements and assuming a comparable (medium) effect size to that estimated in similar studies, an alpha of 0.05 and a minimum of 90% power.

High levels of acceptability and improvements in outcomes (e.g. breast cancer-specific quality of life, anxiety and depressive symptoms, psychological flexibility, self-compassion, health-related costs) are expected at post-treatment and follow-up. This trial seeks to contribute to the integration of brief and cost-effective psychosocial interventions in the usual healthcare for BC patients and survivors.

ELIGIBILITY:
Inclusion Criteria:

- Women with breast cancer who had previously shown interest in participating in the "Mind Programme for Women with Breast Cancer" (original multiple-session version), but were either not eligible or were allocated to the waiting list, and had given permission to be contacted.

Exclusion Criteria:

* current diagnosis of stage IV breast cancer;
* active severe psychopathology (major depression, bipolar disorder, psychotic disorder, substance abuse) or suicidal ideation. These women will follow the standardized procedure in the Portuguese National Health System (SNS) and be referred to psychological and/or psychiatric services for individual and regular support;
* inability to understand and answer to self-report questionnaires in Portuguese;
* no access to a computer, tablet or smartphone with internet.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible participants include females who self-identify as women.
Enrollment: 40 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Quality of life of cancer patients | Baseline (before One-Day Mind Programme) / post-treatment (10 days after One-Day Mind Programme) / 3-month follow-up (3 months after One-Day Mind Programme).
  This outcome will be assessed through the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). EORTC QLQ-C30 comprises 30 items and scores range from 0 to 100 units for each scale and item: 1. Functional Scales: Higher scores indicate better functioning and quality of life; 2. Symptom Scales/Items: Higher scores indicate a higher level of symptoms or problems.
Quality of life of breast cancer patients | Baseline (before One-Day Mind Programme) / post-treatment (10 days after One-Day Mind Programme) / 3-month follow-up (3 months after One-Day Mind Programme).
  This outcome will be assessed through the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Breast Cancer 23 (EORTC QLQ-BR23). EORTC QLQ-BR23 scores range 0 to 100 units for each scale and item: 1. Functional Scales/Items (Body Image, Sexual Functioning, Sexual Enjoyment and Future Perspective): Higher scores indicate better functioning and quality of life; 2. Symptom Scales/Items (Systemic Therapy Side Effects, Breast Symptoms, Arm Symptoms and Upset by Hair Loss): Higher scores indicate a higher level of symptoms or problems.

SECONDARY OUTCOMES:
Depressive symptoms and anxiety severity | Baseline (before One-Day Mind Programme) / post-treatment (10 days after One-Day Mind Programme) / 3-month follow-up (3 months after One-Day Mind Programme).
  This outcome will be assessed through the Hospital Anxiety and Depression Scale (HADS). HADS is a 14-item questionnaire and each item is scored from 0 to 3 units, resulting in subscale scores ranging from 0 to 21 units: 1. Anxiety subscale: Higher scores indicate higher anxiety level; 2. Depression subscale: Higher scores indicate higher depression level.
Psychological flexibility | Baseline (before One-Day Mind Programme) / post-treatment (10 days after One-Day Mind Programme) / 3-month follow-up (3 months after One-Day Mind Programme).
  This outcome will be assessed through the Comprehensive Assessment of Acceptance and Commitment Therapy Processes (CompACT) 18-item version. Each item of CompACT is rated on a scale from 0 to 6, resulting in subscale scores ranging from 0 to 36 units: 1. Openness to Experience subscale: Higher scores indicate more willingness to experience thoughts and feelings without trying to avoid them; 2. Behavioural Awareness subscale: Higher scores indicate more ability to be aware of and engage in behaviours that are consistent with one's values; 3. Valued Action subscale: Higher scores indicate higher extent to which individuals take actions that are aligned with their personal values.
Self-compassion | Baseline (before One-Day Mind Programme) / post-treatment (10 days after One-Day Mind Programme) / 3-month follow-up (3 months after One-Day Mind Programme).
  This outcome will be assessed via Self-Compassion Scale (SELFCS) 26-item version. Each item of SELFCS is rated on a scale from 1 to 5, resulting in subscale scores ranging from 4 or 5 to 20 or 25 units: 1.Self-Kindness subscale(ss): Higher scores indicate higher ability to be kind and understanding towards oneself, especially during difficult times; 2.Self-Judgment ss: Higher scores indicate higher tendency to be overly critical and judgmental of oneself;3.Common Humanity ss: Higher scores indicate higher recognition that suffering and personal failures are part of the shared human experience; 4.Isolation ss: Higher scores indicate higher feelings of isolation and disconnection from others when experiencing suffering; 5.Mindfulness ss: Higher scores indicate higher ability to hold one's painful thoughts and feelings in balanced awareness; 6.Over-Identification ss: Higher scores indicate higher tendency to become overly absorbed and fixated on one's negative emotions and thoughts.
Health-related quality of life | Baseline (before One-Day Mind Programme) / post-treatment (10 days after One-Day Mind Programme) / 3-month follow-up (3 months after One-Day Mind Programme).
  This outcome will be assessed through the EuroQol-5D-5L (EQ-5D-5L). It consists of two main parts: the descriptive system (5 items representing 5 dimensions, that are scored on a scale from 1 to 5 levels of severity: 1. Mobility; 2. Self-care; 3. Usual activities; 4. Pain/Discomfort; 5. Anxiety/Depression) and the EQ visual analogue scale (that records the respondent's self-rated health on a vertical visual analogue scale, where the endpoints are labelled '100 = The best health you can imagine' and '0 = The worst health you can imagine'). Higher scores in both parts indicate higher health-related quality of life and perceived overall health.
Economic impact of cancer on patients | Baseline (before One-Day Mind Programme) / 3-month follow-up (3 months after One-Day Mind Programme).
  This outcome will be assessed through a questionnaire adapted from the UK Cancer Costs Questionnaire (UKCC) Version 2.0. This questionnaire captures the financial burden associated with cancer diagnosis and treatment and has 4 key components: 1. Healthcare Utilization (4 open-ended questions regarding the number of contacts with health professionals outside the hospital setting); 2. Out-of-Pocket Expenses (3 open-ended questions regarding the direct costs incurred by patients, such as medication, travel, and other healthcare-related expenses); 3. Employment and Productivity (5 open-ended questions and 2 multiple-choice questions regarding the impact of cancer on the patient's employment status, including loss of earnings and productivity due to illness); 4. Informal Care (1 open-ended questions regarding the amount of informal care provided by family and friends). Higher scores indicate higher economic impact of cancer and its treatment on patients.
Acceptability of the intervention | At post-treatment (10 days after One-Day Mind Programme).
  This outcome will be assessed through a final evaluation form with 8 items rated on a 5-point Likert scale (1 = Totally Disagree; 5 = Totally Agree) regarding several aspects of the programme (e.g. expectations, satisfaction, usefulness). Higher scores indicate higher acceptance of the intervention by patients.
Feasibility of the intervention: adherence. | Throughout the One-Day Mind Programme (up to 7 hours).
  This outcome will be assessed through direct observation of the patients during the intervention and via attendance records. Higher number of interactions during the intervention and higher attendance indicate higher adherence to the intervention.
Feasibility of the intervention: dropout. | Throughout the One-Day Mind Programme (up to 7 hours).
  This outcome will be assessed via attendance records and it will involve calculating the percentage of patients who discontinue the programme before its completion. A higher percentage will indicate higher dropout rate.

OTHER OUTCOMES:
Impact of significant life events - controlling variable | Baseline (before One-Day Mind Programme) / 3-month follow-up (3 months after One-Day Mind Programme).
  This outcome will be assessed through the Major Life Event Questionnaire (MLEQ). This Portuguese questionnaire comprises 23 items that represent major life events that may occur in a person's life (e.g. marriage, pregnancy, serious illness). For each item, participants are asked to report the occurrence (yes = 1) or absence (no = 0) of the specific event in the previous months (the number of months depends on the moment of assessment). The higher the score (min: 0; max: 23), the higher the number of major life events in the previous months.
Sociodemographic and clinical variables - controlling variable | Baseline (before One-Day Mind Programme).
  This outcome will be assessed through a questionnaire with 47 open-ended or multiple-choice questions regarding sociodemographic (e.g. age) and clinical data (e.g. cancer stage). This data will be important to check inclusion/exclusion criteria.
Psychological processes awareness - planned moderator | Post-treatment (10 days after One-Day Mind Programme).
  This outcome will be assessed through the Awareness of Contextual Therapies Processes Scale (ACTPS). ACTPS is 9-item tool used to measure the processes involved in contextual therapies, such as Acceptance and Commitment Therapy (ACT). Each item is rated on a 5-point Likert scale (1 = Strongly Disagree; 5 = Strongly Agree), resulting in total scores ranging from 9 to 45 units, the higher the score, the higher the awareness level.
Efficacy expectancy - planned moderator | Baseline (before One-Day Mind Programme).
  Yes-no single question about the efficacy expectancy: "Do you believe that the intervention will bring benefits to your quality of life and mental health?"
Home practice frequency - planned moderator | 3-month follow-up (3 months after One-Day Mind Programme).
  Multiple choice question regarding the frequency of home practice in the last 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Research in Neuropsychology and Cognitive and Behavioral Intervention (CINEICC)/Faculty of Psychology and Educational Sciences of the University of Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dinapoli L, Colloca G, Di Capua B, Valentini V. Psychological Aspects to Consider in Breast Cancer Diagnosis and Treatment. Curr Oncol Rep. 2021 Mar 11;23(3):38. doi: 10.1007/s11912-021-01049-3. PMID 33709235
- [Background] Wilkinson L, Gathani T. Understanding breast cancer as a global health concern. Br J Radiol. 2022 Feb 1;95(1130):20211033. doi: 10.1259/bjr.20211033. Epub 2021 Dec 14. PMID 34905391
- [Background] Dochat C, Wooldridge JS, Herbert MS, Lee MW, Afari N. Single-Session Acceptance and Commitment Therapy (ACT) Interventions for Patients with Chronic Health Conditions: A Systematic Review and Meta-Analysis. J Contextual Behav Sci. 2021 Apr;20:52-69. doi: 10.1016/j.jcbs.2021.03.003. Epub 2021 Mar 6. PMID 33868913
- [Background] Trindade IA, Soares A, Skvarc D, Carreiras D, Pereira J, Lourenco O, Sampaio F, de Sousa B, Martins TC, Boaventura P, Marta-Simoes J; Mind Project Team; Moreira H. Efficacy and cost-effectiveness of an ACT and compassion-based intervention for women with breast cancer: study protocol of two randomised controlled trials 1. Trials. 2025 Jan 3;26(1):5. doi: 10.1186/s13063-024-08626-4. PMID 39754194
- [Background] Registo Oncológico Nacional (November, 2023). Registo Oncológico Nacional de Todos os Tumores na População Residente em Portugal, em 2020. https://ron.min-saude.pt/media/2223/ron-2020.pdf
- [Background] Malpus Z, Nazar Z, Smith C, Armitage L. Compassion focused therapy for pain management: '3 systems approach' to understanding why striving and self-criticism are key psychological barriers to regulating activity and improving self-care for people living with persistent pain. Br J Pain. 2023 Feb;17(1):87-102. doi: 10.1177/20494637221133630. Epub 2022 Oct 16. PMID 36815069
- [Background] Gloster, A. T., Walder, N., Levin, M. E., Twohig, M. P., & Karekla, M. (2020). The empirical status of acceptance and commitment therapy: A review of meta-analyses. Journal of Con-textual Behavioral Science, 18, 181-192. https://doi.org/10.1016/j.jcbs.2020.09.009